CLINICAL TRIAL: NCT06257173
Title: The Impact of Patient Safety Education Through Peer Education Model on Patent Safety Competence and Medical Error Attitudes of Student Nurses: A Randomized Controlled Study
Brief Title: Peer Education Impact on Student Nurse Patient Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Miray Aksu, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBU-HEM-MA-01
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nurse-Patient Relations
Keywords: Patient Safety; Medical Errors; Nurse; Students
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This research will be conducted as an experimental study with pretest-posttest randomised control group design.
Who Masked: Participant
Masking Description: Experimental and control groups will be determined using https://www.randomizer.org.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental groups (Experimental): The experimental group will be selected among the students who do not take the "Patient and Employee Safety" course and who volunteer to participate in the study.The experimental group will receive 2 hours of patient safety training with a peer educator. Data collection forms will be applied at the end of the training, and data collection forms will be applied again 6 weeks after the training.
  Interventions: Behavioral: Education
- Control groups (No Intervention): The control group will be selected among the students taking the "Patient and Employee Safety" course who volunteer to participate in the studyThe control group will be given 2 hours of patient safety training in the curriculum by the researcher. Data collection forms will be applied at the end of the training, and data collection forms will be applied again 6 weeks after the training.

INTERVENTIONS:
Behavioral: Education — The experimental group will receive 2 hours of patient safety training with a peer educator.
  Arms: Experimental groups

SUMMARY:
The World Health Organisation (WHO) and the Ministry of Health define patient safety as the prevention of errors and adverse effects. Medical errors are a global problem and one out of every 10 patients is seriously harmed. The importance of education and attitudes of health personnel for patient safety is emphasised. Providing patient safety education to nursing students is important to provide quality health care. Peer education model stands out as an effective method to increase the patient safety competence of students. The study was planned as a randomised controlled study to evaluate the effect of patient safety education given according to the peer education model on the patient safety competence of student nurses and their attitudes towards medical errors.

DETAILED DESCRIPTION:
The World Health Organisation (WHO) defines patient safety as "the prevention of errors related to health services and negative effects on patients". In our country, within the scope of the Ministry of Health Quality Standards in Health, patient safety is defined as "measures and improvement activities that can be taken to keep all foreseeable hazards that may cause harm to all stakeholders receiving services at an acceptable level of risk".Patient safety is a global problem that concerns many countries around the world. This problem stems from the large number of reported patient outcomes related to medical errors . Medical errors can cause permanent injuries and prolonged hospital stays and even death in patients. According to the World Health Organisation, one in 10 patients is seriously harmed by medical errors. Prevention of medical errors and their effects is the main goal of patient safety. ICN has stated that in order to increase patient safety, comprehensive measures should be taken in recruitment, training and retention of professional health care personnel, fight against infection, safe use of drugs, improvement of their performance, device safety, healthy practice and care environment, environmental safety and risk management, and scientific knowledge on patient safety and the infrastructure that will enable its development should be combined as a whole.

It is the responsibility of all healthcare professionals to prevent and prevent medical errors and to ensure patient safety. In this context, considering the time nurses spend with patients, it is also indispensable for nursing care. For this reason, it is of great importance to determine the attitudes of health professionals in medical errors in order to reduce medical error rates, thus ensuring patient safety and increasing trust in health institutions.

Medical errors caused by healthcare professionals are preventable errors, and patient safety can be ensured by creating an effective and strong patient safety culture through trainings. Medical errors and risks can be minimised by establishing and developing a patient safety culture and adopting it by all healthcare professionals and future healthcare professionals (students). It is very important to educate nursing students, who will be the health professionals of the future, about patient safety in order to provide safe and quality health care. Encountering a new patient in the practice area and performing any application to this patient for the first time may cause anxiety and fear in students, which may lead students to make medical errors. Teaching the basic concept of patient safety through patient safety education in nursing undergraduate programmes is an important step towards ensuring patient safety and quality in clinical practice, in addition to helping nursing students see the "big picture" for safer care and to have a good knowledge of basic principles before providing nursing care in the clinical field.

Nursing students in recent years are more present in clinics and learn how to communicate with patients and work with other health professionals, which can increase their patient safety competence. To effectively improve student patient safety competence, it is necessary to develop and implement a range of teaching methods such as clinical practice as well as laboratory/simulation sessions . It is also recommended to create actionable strategies that bring together administrators, educators, students and patients to coordinate teaching with the clinic by evaluating whether there is a change in students' knowledge, skills and behaviours in quality and patient safety with objective methods. In line with these recommendations, it is very important that the courses given in undergraduate education are given with an innovative approach to increase patient safety and quality of care.

One of the effective educational methods that facilitate health promotion and create an appropriate learning environment is peer education. A peer is an individual who belongs to the same social group as the learner and is believed to have similar abilities to the learner and can act as a strong motivator in learning. Peers can communicate better, share their experiences and encourage each other to adopt appropriate health behaviours. Peer teaching, an effective educational approach for nursing students, is based on Bandura's social learning theory, which assumes that learning alone restricts the person to observe the attitudes of others. Recently, the peer education model has been proposed as an alternative to traditional educational approaches as it is recognised to have many advantages.

The success of the peer education model is closely related to the fact that peers support each other, express themselves more comfortably, perform their skills that they cannot reveal under the supervision of an authority more easily, and learn less stressful. From this point of view, it is expected that the patient safety education to be given to nursing students using the peer education module will contribute positively to students' patient safety competence and attitudes towards medical errors. In addition, it is thought to contribute to the studies examining the effect of patient safety education, which is limited in the literature. The study was planned as a randomised controlled study to evaluate the effect of patient safety education given according to the peer education model on student nurses' patient safety competence and attitudes towards medical errors.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* To be a 3rd year student of SBÜ Gülhane Faculty of Nursing in 2023-2024 academic year
* No visual or hearing impairment

Exclusion Criteria:

* Voluntary withdrawal from the research
* Not participating in the research phases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Patient Safety Competency Self-Assessment Tool | six weeks
  The Patient Safety Competency Self-Assessment Tool consists of 41 items in three dimensions: knowledge (six items), skills (21 items) and attitudes (14 items). The total mean scores of the instrument and each of the three subscales range from one to five, with higher scores indicating higher overall competence and competence in knowledge, skills and attitudes.
Attitude Scale on Medical Errors | six weeks
  The Attitude Towards Medical Errors Scale (ATMS) consists of 16 items and 3 subscales (medical error perception, medical error approach, and reasons for medical errors). The 10th and 13th items are reverse scored. In the scale calculation, the scale total score is taken and the scale score is obtained by dividing the raw score obtained by the number of scale items. In the sub-dimension score calculation, the sub-dimension score is totalled and divided by the number of sub-dimension items. is divided and the score obtained is evaluated between 1-5. The cut-off point of the scale was determined as 3. Medical error attitudes of those who score below 3 on the scale are evaluated as negative, and medical error attitudes of those who score 3 and above are evaluated as positive.

SECONDARY OUTCOMES:
The Descriptive Information Form | six weeks
  The Introductory Information Form is a form consisting of 8 questions designed by the researchers to define the students' age, gender, reason for choosing the profession, status of receiving education on patient safety, patient safety education and knowledge about medical errors.

CONTACTS AND LOCATIONS:
Overall Officials: Miray Aksu, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No